CLINICAL TRIAL: NCT02546856
Title: Safety and Effectiveness of Drug up Titration by Nurses Specialized in Heart Failure (HF) Patients
Acronym: ETIFIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Collaborators: Carlos III Health Institute (Other Government); Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Maria Juana Oyanguren Artola, Heart Failure Nurse, Hospital Galdakao-Usansolo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PI14/01208
Record Dates: First submitted 2015-05-18; First posted 2015-09-11 (Estimated); Results first posted 2020-11-27 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Heart Failure
Keywords: Up-titration; Nursing or Nurse; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heart Failure (HF) cardiologist up-titration (Active Comparator): Active Comparator:Cardiologist decides dosage with nursing clinical and educational support.
  Interventions: Other: Heart Failure (HF) cardiologist up-titration
- HF nurse up-titration (Experimental): Intervention: The cardiologist prescribes drugs and, driven by protocol, the HF nurse implements the up-titration.
  Interventions: Other: Heart Failure (HF) nurse up-titration

INTERVENTIONS:
Other: Heart Failure (HF) nurse up-titration — Up-titration of Beta-Blocker (BB), Angiotensin Converting Enzyme Inhibitor (ACEI), Angiotensin II Receptor Blocker (ARB) and Mineralocorticoid Receptor Antagonist (MRA) in Heart Failure "De Novo" patients with Left Ventricular Ejection Fraction (LVEF)≤ 40%, following a protocol based on 2012 European Society of Cardiology (ESC) Heart Failure (HF) guidelines with cardiologist prescription and support.
  Arms: HF nurse up-titration
Other: Heart Failure (HF) cardiologist up-titration — Up-titration of Beta-Blocker (BB), Angiotensin Converting Enzyme Inhibitor (ACEI), Angiotensin II Receptor Blocker (ARB) and Mineralocorticoid Receptor Antagonist (MRA) in Heart Failure "De Novo" patients with Left Ventricular Ejection Fraction (LVEF)≤ 40%, following a protocol based on 2012 European Society of Cardiology (ESC) Heart Failure (HF) guidelines. Drugs are prescribed and titrated by the cardiologist.
  Arms: Heart Failure (HF) cardiologist up-titration

SUMMARY:
Introduction: Heart Failure (HF) generates multiple hospital admissions and mortality, which are reduced with the administration of Beta-Blocker (BB), Angiotensin Converting Enzyme Inhibitor (ACEI), Angiotensin II Receptor Blocker (ARB) and Mineralocorticoid Receptor Antagonist (MRA) drugs (Level of Evidence A). The effect is dose-dependent. Nevertheless, dosages are suboptimal. European Guidelines 2012 recommend close monitoring and up-titration of drugs by HF nurses. Trials are needed to evaluate their effectiveness and safety. Objective: To compare doses achieved by patients of BB, ACEI, ARB II and MRA in 4 months ( % relative to target doses) in the intervention group (HF nurse) and in the control group ( cardiologist), adverse events, Left Ventricular Ejection Fraction (LVEF), New York Heart Association (NYHA), 6 min. walking test, quality of life, Nt-proBNP, readmissions and mortality. Hypothesis: Non-inferiority. Design: Multicenter randomized controlled trial. New ("de novo") HF patients with LVEF ≤ 40%, NYHA II-III, without contraindications to BB of 17 Spanish hospitals will be included. Intervention: The cardiologist prescribes drugs and, driven by protocol, the HF nurse implements the up-titration. In the control group doses are decided by the cardiologist clinical support and education being provided by nurses. Variables: age, sex, education, psycho-social level, Cardio Vascular Risk Factors (CVRF), NYHA, LVEF, ischemic cardiopathy., N-terminal pro B-type natriuretic peptide (Nt-proBNP), 6min. walking test, Creatinine/Glomerular Filtration Rate (GFR), Potassium (K), haemoglobin, Blood Pressure (BP), Heart Rate (HR), mg./drug, European Heart Failure Self-Care Behaviour Scale (EHFScBS), Minnesota Living with Heart Failure questionnaire (MLHFQ), European Quality of life Scale (EQ-5D). Expected Results: If our hypothesis were confirmed, evidence would be provided on the effectiveness of this healthcare management, that could be economically evaluated in future studies. A qualitative study also will be undertaken to explore barriers and facilitators to implementation

DETAILED DESCRIPTION:
No apply

ELIGIBILITY:
Inclusion Criteria:

* Patient with "de novo" heart Failure and LVEF <= 40% admitted in hospital, without contraindications for BB prescription with cardiologist up-titration prescription and without having achieved BB target dose previous discharge and signing informed consent.

Exclusion Criteria:

* Contraindications for BB.
* Living in a nursing home.
* Life expectancy < 6 months.
* Unable to self-care or mental disease without caregiver.
* Unable to weight
* Without phone
* Unable to go to clinic visit.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2015-03; Primary Completion 2018-10 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Juana Oyanguren, Nurse, Principal Investigator — Osakidetza-Servicio vasco de Salud
Locations (1):
- Hospital de usansolo-Galdakao, Usansolo, Bizkaia, Spain

REFERENCES:
- [Background] Oyanguren J, Garcia-Garrido L, Nebot Margalef M, Lekuona I, Comin-Colet J, Manito N, Roure J, Ruiz Rodriguez P, Enjuanes C, Latorre P, Torcal Laguna J, Garcia-Gutierrez S; ETIFIC7 research group. Design of a multicentre randomized controlled trial to assess the safety and efficacy of dose titration by specialized nurses in patients with heart failure. ETIFIC study protocol. ESC Heart Fail. 2017 Nov;4(4):507-519. doi: 10.1002/ehf2.12152. Epub 2017 Apr 3. PMID 29154427
- [Result] Oyanguren J, Garcia-Garrido L, Nebot-Margalef M, Latorre-Garcia P, Torcal-Laguna J, Comin-Colet J, Roure J, Gonzalez-Costello J, Manito N, Garcia-Pinilla JM, Sanchez-Paule Y, Varela-Roman A, Moure M, Segovia-Cubero J, Soria T, Arana-Arri E, Lekuona I; Steering Committee on behalf of the ETIFIC research team group. Noninferiority of heart failure nurse titration versus heart failure cardiologist titration. ETIFIC multicenter randomized trial. Rev Esp Cardiol (Engl Ed). 2021 Jun;74(6):533-543. doi: 10.1016/j.rec.2020.04.016. Epub 2020 Jun 24. English, Spanish. PMID 32591295
- [Derived] Oyanguren J, Diaz-Molina B, Lekuona I, Gonzalez-Costello J, Lopez-Fernandez S, Garcia-Pinilla JM, Garcia-Garrido L, Lopez-Moyano G, Manito N, Cobo-Marcos M, Nebot-Margalef M, Latorre-Garcia P, Arana-Arri E, Perez-Fernandez S, Torcal-Laguna J; ETIFIC research team group. Gender differences in drug titration among heart failure patients with reduced ejection fraction in the ETIFIC trial. Rev Esp Cardiol (Engl Ed). 2022 Aug;75(8):636-648. doi: 10.1016/j.rec.2021.11.002. Epub 2021 Dec 10. English, Spanish. PMID 34903479

RESULTS

PARTICIPANT FLOW:
Groups:
- Heart Failure (HF) Nurse Up-titration: Intervention:The cardiologist prescribes drugs and the HF-nurse implements the up-titration, driven by protocol based on 2012 ESC HF guidelines, with cardiologist support.
  Up-titration of Beta-Blocker (BB), Angiotensin Converting Enzyme Inhibitor (ACEI), Angiotensin II Receptor Blocker (ARB) and Mineralocorticoid Receptor Antagonist (MRA) drugs of Heart Failure "De Novo" Left Ventricular Ejection Fraction ≤ 40% Patients
- Heart Failure (HF) Cardiologist Up-titration: Active Comparator:The cardiologist prescribes and decides dosage following a protocol based on 2012 ESC HF guidelines, with nursing clinical and educational support.
  Up-titration of Beta-Blocker (BB), Angiotensin Converting Enzyme Inhibitor (ACEI), Angiotensin II Receptor Blocker (ARB) and Mineralocorticoid Receptor Antagonist (MRA) drugs of Heart Failure "De Novo" Left Ventricular Ejection Fraction ≤ 40% Patients
Period: 4 Months Evaluation
Arm/Group | Heart Failure (HF) Nurse Up-titration | Heart Failure (HF) Cardiologist Up-titration
Started | 164 | 156
Completed | 144 | 145
Not Completed | 20 | 11
Not completed — Death | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 3 | 3
Not completed — Physician Decision | 3 | 0
Not completed — Working or living abroad | 5 | 1
Not completed — reasons not due to titration | 4 | 1
Not completed — HF Unit not active in summer | 1 | 0
Period: 6 Months Evaluation
Arm/Group | Heart Failure (HF) Nurse Up-titration | Heart Failure (HF) Cardiologist Up-titration
Started | 144 | 145
Completed | 136 | 138
Not Completed | 8 | 7
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Working or living abroad | 6 | 4
Not completed — reasons not due to titration | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Heart Failure (HF) Cardiologist Up-titration: Active Comparator:Cardiologist decides dosage with nursing clinical and educational support.
  HF cardiologist up-titration: Up-titration of Beta-Blocker (BB) in Heart Failure " De Novo" Left Ventricular Ejection Fraction ≤ 40% Patients, following a protocol based on 2012 ESC HF guidelines
  HF cardiologist up-titration: Up-titration of Angiotensin Converting Enzyme Inhibitor (ACEI) in Heart Failure " De Novo" Left Ventricular Ejection Fraction ≤ 40% Patients, following a protocol based on 2012 ESC HF guidelines
  HF cardiologist up-titration: Up-titration of Angiotensin II Receptor Blocker (ARB) in Heart Failure " De Novo" Left Ventricular Ejection Fraction≤ 40% Patients, following a protocol based on 2012 ESC HF guidelines
  HF cardiologist up-titration: Up-titration of Mineralocorticoid Receptor Antagonist (MRA) in Heart Failure " De Novo" Left Ventricular Ejection Fraction ≤ 40% Patients, following a protocol based on 2012 ESC HF guidelines
- HF Nurse Up-titration: Patients, following a protocol based on 2012 ESC HF guidelines. Cardiologist prescription and support
  HF nurse up-titration: Up-titration of Beta-Blocker (BB) in Heart Failure " De Novo" Left Ventricular Ejection Fraction ≤ 40% Patients, following a protocol based on 2012 ESC HF guidelines.
  HF nurse up-titration: Up-titration of Angiotensin Converting Enzyme Inhibitor (ACEI) in Heart Failure " De Novo" Left Ventricular Ejection Fraction ≤ 40% Patients, following a protocol based on 2012 ESC HF guidelines.
  HF nurse up-titration: Up-titration of Angiotensin II Receptor Blocker (ARB) in Heart Failure " De Novo" Left Ventricular Ejection Fraction ≤ 40% Patients. Protocol based on 2012 ESC HF guidelines.
  HF nurse up-titration: Up-titration of Mineralocorticoid Receptor Antagonist (MRA) in Heart Failure " De Novo" Left Ventricular Ejection Fraction ≤ 40% Patients, . Protocol based on 2012 ESC HF guidelines.
- Total: Total of all reporting groups
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration | Total
Number analyzed (Participants) | 156 | 164 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.64 (12.25) | 61.88 (12.14) | 61.28 (12.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 45 | 83
  Male | 118 | 119 | 237
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 156 | 164 | 320
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 156 | 164 | 320
betablocker mean relative dose [Mean (Standard Deviation); unit: % to target dose] — betablocker mean relative dose ( % to target dose) at baseline Population: n considered for baseline doses In both groups: patients, who were at the time of measuring the achieved doses after titration, the 4th month. We evaluated the 4 month titration process made by HF cardiologist vs HF nurse. Patients who left the study did not receive this intervention.
  % to target dose
    number analyzed (Participants) | 145 | 144 | 289
    (all) | 34.80 (20.6) | 34.81 (18.16) | 34.80 (19.38)
left ventricular ejection fraction % [Mean (Standard Deviation); unit: %of blood leaving the heart /beat] — Ejection fraction is a measurement of the percentage of blood leaving the heart each time it contracts.
  %of blood leaving the heart /beat | 27.45 (7.25) | 27.95 (6.69) | 27.71 (6.97)
Nt-proBNP [Mean (Standard Deviation); unit: pg/ml] — Nt-proBNP (N-terminal pro-B type natriuretic peptide) at discharge mean (SD) Population: other patients had BNP
  pg/ml
    number analyzed (Participants) | 139 | 145 | 284
    (all) | 3001 (4041) | 3425 (5256) | 3217 (4697)
6 minute walking test [Mean (Standard Deviation); unit: meters] — 6 minute walking test, meters. Six minute walking test. Measurement of exercise capacity . It provides information regarding functional capacity, response to therapy and prognosis across a range of chronic cardiopulmonary conditions. The six-minute walk test (6MWT) measures the distance (meters) an individual is able to walk over a total of six minutes on a hard, flat surface.
  meters | 370 (108) | 361 (102) | 366 (105)
Number of participants with New York Heart Association (NYHA) I,II,III,IV [Count of Participants; unit: Participants] — Number of participants class I-IV New York Heart Association (NYHA) functional classification based on severity of symptoms and physical activity:
  NYHA I (better): No limitation of physical activity NYHA II: Slight limitation of ordinary physical activity, breathlessness NYHA III: marked limitation of physical activity. Comfortable at rest, but less than ordinary activity results in undue breathlessness, fatigue or palpitations NYHA IV ( worse): unable to carry on any physical activity without discomfort.Symptoms at rest can be present. If any physical activity, discomfort is increased.
  Participants
    NYHA I | 0 | 0 | 0
    NYHA II | 128 | 139 | 267
    NYHA III | 28 | 25 | 53
    NYHA IV | 0 | 0 | 0
Minnesota living with heart failure questionnaire [Mean (Standard Deviation); unit: units on a scale] — Quality of Life measured by Minnesota Living With Heart Failure Questionnaire (MLWHFQ). The content of this questionnaire was selected to be representative of the ways heart failure and treatments can affect the key physical, emotional, social and mental dimensions of quality of life of patients with heart failure. It consist of 21-items with score 0-5. Final evaluation moves from 0 (none) to 105 (very much); a lower score means better quality of life.
  units on a scale | 45.71 (22.21) | 50.8 (22.61) | 48.31 (22.52)
European Quality of Life Scale: EuroQol- 5 Dimension index [Mean (Standard Deviation); unit: score on a scale] — European Quality of Life Scale: EuroQol- 5 Dimension index (Range: 1 full health-0 death). It measures health status self-reported by the patient. It has 5 domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is divided into three levels: 1 no problem; 2 moderate problems; 3 extreme problems. This information is converted into a single summary index, by applying a formula that attaches specific country values to each of the levels in each dimension, that are subtracted from 1 (the full health). EQ-5D-3L-User-Guide_version-6.0 (1).pdf
  score on a scale | 0.75 (0.24) | 0.73 (0.23) | 0.74 (0.23)
ACEI mean relative dose [Mean (Standard Deviation); unit: % to target dose] — angiotensin-converting enzyme inhibitors mean relative dose ( % to target dose described in european heart failure guidelines) Population: n considered to calculate the mean baseline doses of ACEI in both groups: only the patients who received a prescription at baseline were included in the analysis.
  Every patient was prescribed betablocker but not ACEI. Alternatively It was possible to be prescribed ARB/sacubitril-valsartan or nothing
  % to target dose
    number analyzed (Participants) | 121 | 118 | 239
    (all) | 40.13 (25.38) | 45.92 (30.06) | 43.04 (27.81)
Angiotensin II Receptor Blockers (ARB) mean relative dose [Mean (Standard Deviation); unit: % to target dose] — ARB, angiotensin II receptor blockers, mean relative dose ( % to target dose).Target dose is described in European guidelines. Measured at baseline. Population: n considered to calculate the mean baseline doses of ARA in both groups: only the patients who received a prescription at baseline were included in the analysis.
  Every patient was prescribed betablocker but not ARB. Alternatively It was possible to be prescribed ACEI/sacubitril-valsartan or nothing
  % to target dose
    number analyzed (Participants) | 8 | 16 | 24
    (all) | 43.20 (20.63) | 29.15 (14.99) | 33.84 (17.95)
MRA mean relative dose [Mean (Standard Deviation); unit: % to target dose] — mineralocorticoid-receptor antagonists mean relative dose (% to target dose described in european heart failure guidelines) Population: n for MRA baseline doses in both groups: patients, who were at the time of measuring the achieved doses after titration, the 4th month and had a prescription during the titration period at any time.
  Every patient was prescribed betablocker but not MRA. It was possible not having the need of its prescription.
  % to target dose
    number analyzed (Participants) | 127 | 125 | 252
    (all) | 63.18 (33.00) | 61.4 (33.52) | 62.30 (33.21)

OUTCOME MEASURES:

1. Primary Outcome: BB % Relative Dose (Mean) With Regard to Target Dose
Description: BB mean Relative dose is the mean dose of betablockers achieved 4 months after starting titration, relative to target dose ( %) , which is the target dose of european heart failure guidelines for BB.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: percentage of target dose
Groups:
- Heart Failure (HF) Cardiologist Up-titration: Active Comparator:Cardiologist decides dosage with nursing clinical and educational support.
  HF cardiologist up-titration: Up-titration of Beta-Blocker (BB) in Heart Failure " De Novo" Left Ventricular ejection Fraction ≤ 40% Patients, following a protocol based on 2012 ESC HF guidelines
  HF cardiologist up-titration: Up-titration of Angiotensin Converting Enzyme Inhibitor (ACEI) in Heart Failure " De Novo" Left Ventricular ejection Fraction ≤ 40% Patients, following a protocol based on 2012 ESC HF guidelines
  HF cardiologist up-titration: Up-titration of Angiotensin II Receptor Blocker (ARB) in Heart Failure " De Novo" Left Ventricular ejection Fraction ≤ 40% Patients, following a protocol based on 2012 ESC HF guidelines
  HF cardiologist up-titration: Up-titration of Mineralocorticoid Receptor Antagonist (MRA) in Heart Failure " De Novo" Left Ventricular ejection Fraction ≤ 40% Patients, following a protocol based on 2012 ESC HF guidelines
- HF Nurse Up-titration: Intervention: The cardiologist prescribes drugs and, driven by protocol, the HF nurse implements the up-titration.
  HF nurse up-titration: Up-titration of Beta-Blocker (BB) in Heart Failure " De Novo" Left Ventricular ejection Fraction (EF) ≤ 40% Patients. Protocol based on 2012 European Society of Cardiology (ESC) HF guidelines.
  HF nurse up-titration: Up-titration of Angiotensin Converting Enzyme Inhibitor (ACEI) in Heart Failure " De Novo" EF≤ 40% Patients. Protocol based on 2012 ESC HF guidelines.
  HF nurse up-titration: Up-titration of Angiotensin II Receptor Blocker (ARB) in Heart Failure " De Novo" EF≤ 40% Patients. Protocol based on 2012 ESC HF guidelines.
  HF nurse up-titration: Up-titration of Mineralocorticoid Receptor Antagonist (MRA) in Heart Failure " De Novo" EF≤ 40% Patients. Protocol based on 2012 ESC HF guidelines.
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 145 | 144
percentage of target dose | 56.29 (31.3) | 71.09 (31.05)
Statistical Analysis 1: Comparison: Heart Failure (HF) Cardiologist Up-titration vs HF Nurse Up-titration; Test type: Non-Inferiority — For the hypothesis that the relative dose of BBs would reach 52% by the end of the study and using an equivalence margin of 7%, we would need 157 patients per group for an alpha level of significance of 0.05 and a statistical power of 80% (beta of 0.80); p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 14.8, 95% CI 2-sided [7.5 to 22.1]

2. Secondary Outcome: Number of Participants With Worsening Renal Function (From Baseline to 4th Month)
Description: Number of participants with worsening renal function during the titration process (from baseline to 4 month) that could be associated to the titration process (Creatinine increase >50% baseline creatinine or creatinine>3mg/dl, or Estimated Glomerular Filtration<25 ml/min/1.73 m2)
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Groups:
- Heart Failure (HF) Cardiologist Up-titration: Active Comparator:Cardiologist decides dosage with nursing clinical and educational support.
  HF cardiologist up-titration: Up-titration of Beta-Blocker (BB) in Heart Failure " De Novo" EF≤ 40% Patients, following a protocol based on 2012 ESC HF guidelines
  HF cardiologist up-titration: Up-titration of Angiotensin Converting Enzyme Inhibitor (ACEI) in Heart Failure " De Novo" EF≤ 40% Patients, following a protocol based on 2012 ESC HF guidelines
  HF cardiologist up-titration: Up-titration of Angiotensin II Receptor Blocker (ARB) in Heart Failure " De Novo" EF≤ 40% Patients, following a protocol based on 2012 ESC HF guidelines
  HF cardiologist up-titration: Up-titration of Mineralocorticoid Receptor Antagonist (MRA) in Heart Failure " De Novo" EF≤ 40% Patients, following a protocol based on 2012 ESC HF guidelines
- HF Nurse Up-titration: Intervention: The cardiologist prescribes drugs and, driven by protocol, the HF nurse implements the up-titration.
  HF nurse up-titration: Up-titration of Beta-Blocker (BB) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 European Society of Cardiology (ESC) HF guidelines.
  HF nurse up-titration: Up-titration of Angiotensin Converting Enzyme Inhibitor (ACEI) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 ESC HF guidelines.
  HF nurse up-titration: Up-titration of Angiotensin II Receptor Blocker (ARB) in Heart Failure " De Novo" EF≤ 40% Patients, following a protocol based on 2012 ESC HF guidelines.
  HF nurse up-titration: Up-titration of Mineralocorticoid Receptor Antagonist (MRA) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 ESC HF guidelines.
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 145 | 144
Participants | 6 | 4
Statistical Analysis 1: Comparison: Heart Failure (HF) Cardiologist Up-titration vs HF Nurse Up-titration; Test type: Equivalence — equivalence margin of 5%; p = 0.52, Chi-squared; Difference in percentages = 1.4, 95% CI 2-sided [-3.33 to 6.32]

3. Secondary Outcome: Number of Participants With Potassium (K) ≥5.5 Meq/l (From Baseline to 4 Month)
Description: Number of participants with Potassium≥ 5.5 meq/l during the titration process (from baseline to 4 month) that could be associated to this titration process
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Groups:
- HF Nurse Up-titration: Intervention: The cardiologist prescribes drugs and, driven by protocol, the HF nurse implements the up-titration.
  HF nurse up-titration: Up-titration of Beta-Blocker (BB) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 European Society of Cardiology (ESC) HF guidelines. Cardiologist prescription and support
  HF nurse up-titration: Up-titration of Angiotensin Converting Enzyme Inhibitor (ACEI) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 ESC HF guidelines. Cardiologist prescription and support
  HF nurse up-titration: Up-titration of Angiotensin II Receptor Blocker (ARB) in Heart Failure " De Novo" EF≤ 40% Patients. Protocol based on 2012 ESC HF guidelines. Cardiologist prescription and support
  HF nurse up-titration: Up-titration of Mineralocorticoid Receptor Antagonist (MRA) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 ESC HF guidelines. Cardiologist prescription and support
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 145 | 144
Participants | 3 | 6
Statistical Analysis 1: Comparison: Heart Failure (HF) Cardiologist Up-titration vs HF Nurse Up-titration; Test type: Non-Inferiority — Equivalence margin of 5%; p = 0.31, Chi-squared; Difference in percentages = 2.10, 95% CI 2-sided [-1.9 to 6.1]

4. Secondary Outcome: Number of Participants With Symptomatic Hypotension (From Baseline to 4 Month)
Description: Description: Number of participants with symptomatic hypotension during the titration process (from baseline to 4 month) that could be associated to this titration process. Symptomatic hypotension defined as symptoms such as dizziness or light headedness, associated to hypotension
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 145 | 144
Participants | 13 | 12
Statistical Analysis 1: Comparison: Heart Failure (HF) Cardiologist Up-titration vs HF Nurse Up-titration; Test type: Non-Inferiority — Equivalence margin of 5%; p = 0.85, Chi-squared; Difference in percentages = -0.63, 95% CI 2-sided [-7.1 to 5.85]

5. Secondary Outcome: Number of Participants With Heart Rate (HR) < 50 Beats Per Minute (From Baseline to 4 Month)
Description: Number of participants with Heart Rate (HR) < 50 beats per minute during the titration process (from baseline to 4 month) , which could be associated to the titration process. (with or without symptoms)
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Groups:
- HF Nurse Up-titration: Intervention: The cardiologist prescribes drugs and, driven by protocol, the HF nurse implements the up-titration.
  HF nurse up-titration: Up-titration of Beta-Blocker (BB) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 European Society of Cardiology (ESC) HF guidelines. Cardiologist prescription and support
  HF nurse up-titration: Up-titration of Angiotensin Converting Enzyme Inhibitor (ACEI) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 ESC HF guidelines with cardiologist prescription and support.
  HF nurse up-titration: Up-titration of Angiotensin II Receptor Blocker (ARB) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 ESC HF guidelines. Cardiologist prescription and support
  HF nurse up-titration: Up-titration of Mineralocorticoid Receptor Antagonist (MRA) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 ESC HF guidelines. Cardiologist prescription and support
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 145 | 144
Participants | 7 | 10
Statistical Analysis 1: Comparison: Heart Failure (HF) Cardiologist Up-titration vs HF Nurse Up-titration; Test type: Non-Inferiority — Equivalence margin of 5%; p = 0.44, Chi-squared; Difference in percentages = 2.12, 95% CI 2-sided [-3.3 to 7.54]

6. Secondary Outcome: Number of Patients With Atrio Ventricular (AV) Block Due to Titration
Description: Number of patients with AV Block during the titration process, associated to the BB titration
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Groups:
- HF Nurse Up-titration: Intervention: The cardiologist prescribes drugs and, driven by protocol, the HF nurse implements the up-titration.
  HF nurse up-titration: Up-titration of Beta-Blocker (BB) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 European Society of Cardiology (ESC) HF guidelines. Cardiologist prescription and support
  HF nurse up-titration: Up-titration of Angiotensin Converting Enzyme Inhibitor (ACEI) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 ESC HF guidelines. Cardiologist prescription and support
  HF nurse up-titration: Up-titration of Angiotensin II Receptor Blocker (ARB) in Heart Failure " De Novo" EF≤ 40% Patients. Protocol based on 2012 ESC HF guidelines. Cardiologist prescription and support
  HF nurse up-titration: Up-titration of Mineralocorticoid Receptor Antagonist (MRA) in Heart Failure " De Novo" EF≤ 40% patients,. Protocol based on 2012 ESC HF guidelines. Cardiologist prescription and support
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 145 | 144
Participants | 0 | 0

7. Secondary Outcome: Number of Patients With Worsening of Heart Failure Signs and Symptoms
Description: Number of patients with worsening of heart failure signs and symptoms during the titration process ( from baseline to 4 month) which could be associated to the titration process.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Groups:
- HF Nurse Up-titration: Intervention: The cardiologist prescribes drugs and, driven by protocol, the HF nurse implements the up-titration.
  HF nurse up-titration: Up-titration of Beta-Blocker (BB) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 European Society of Cardiology (ESC) HF guidelines.
  HF nurse up-titration: Up-titration of Angiotensin Converting Enzyme Inhibitor (ACEI) in Heart Failure " De Novo" EF≤ 40% Patients. Protocol based on 2012 ESC HF guidelines.
  HF nurse up-titration: Up-titration of Angiotensin II Receptor Blocker (ARB) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 ESC HF guidelines.
  HF nurse up-titration: Up-titration of Mineralocorticoid Receptor Antagonist (MRA) in Heart Failure " De Novo" EF≤ 40% patients,. Protocol based on 2012 ESC HF guidelines.
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 145 | 144
Participants | 1 | 2
Statistical Analysis 1: Comparison: Heart Failure (HF) Cardiologist Up-titration vs HF Nurse Up-titration; Test type: Non-Inferiority — equivalence margin of 5%; p = 0.56, Chi-squared; Difference in percentages = 0.70, 95% CI 2-sided [-1.6 to 3.04]

8. Secondary Outcome: Number of Patients With Admissions Due to Titration
Description: Number of patients with admissions due to titration ( not due to other causes)
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Groups:
- HF Nurse Up-titration: Intervention: The cardiologist prescribes drugs and, driven by protocol, the HF nurse implements the up-titration.
  HF nurse up-titration: Up-titration of Beta-Blocker (BB) in Heart Failure " De Novo" EF≤ 40% Patient. Protocol based on 2012 European Society of Cardiology (ESC) HF guidelines. Cardiologist prescription and support
  HF nurse up-titration: Up-titration of Angiotensin Converting Enzyme Inhibitor (ACEI) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 ESC HF guidelines. Cardiologist prescription and support
  HF nurse up-titration: Up-titration of Angiotensin II Receptor Blocker (ARB) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 ESC HF guidelines. Cardiologist prescription and support
  HF nurse up-titration: Up-titration of Mineralocorticoid Receptor Antagonist (MRA) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 ESC HF guidelines. Cardiologist prescription and support
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 145 | 144
Participants | 0 | 0

9. Secondary Outcome: Number of Patients: Mortality Due to Titration
Description: Number of patients: Mortality due to titration ( not due to other causes)
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 145 | 144
Participants | 0 | 0

10. Secondary Outcome: Number of Paticipants With Drug Stop (Some Titration Drug Withdrawal Due to Intolerance, no Need or Change to Other Treatment)
Description: number of paticipants with drug Stop ( withdrawal) that occur during the titration process that could be due to an adverse event. ( it can be not only due to an adverse event but because there is no need of this drug or its substitution for another kind of drug)
Time Frame: 4 months
Population: Participants analyzed are only participants with drug withdrawal
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 12 | 9
Participants
  betablocker stop | 3 | 1
  ACEI stop | 3 | 0
  ARB stop | 0 | 1
  MRA stop | 6 | 7

11. Secondary Outcome: Change in % Left Ventricular Ejection Fraction
Description: Change in % Left Ventricular Ejection Fraction (difference of change from baseline to 6 months between groups) Ejection fraction is a measurement of the percentage of blood leaving the heart each time it contracts.
Time Frame: 6 months
Population: It has to be taken into account that in outcome mesasures the order of groups and their number of participants is reversed ( first HF cardiologist, second HF nurse) in regard to those in the participant flow. ( first HF nurse, second HF cardiologist)
Measure: Mean (Standard Deviation); unit: percentage of blood expelled/each beat
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 138 | 136
percentage of blood expelled/each beat | 15.46 (11.46) | 15.63 (13.29)
Statistical Analysis 1: Comparison: Heart Failure (HF) Cardiologist Up-titration vs HF Nurse Up-titration; Test type: Non-Inferiority — Equivalence margin of 5%; p = 0.96, t-test, 2 sided; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-2.69 to 2.83]

12. Secondary Outcome: N-terminal Pro-B Type Natriuretic Peptide Improvement (Nt-proBNP)
Description: Nt-proBNP (N-terminal pro-B type natriuretic peptide) Improvement (Decrease) difference of change from baseline to 6 months between groups, mean (SD)
Time Frame: 6 months
Population: BNP was analysed in 11 patients of both groups, instead of Nt proBNP ( 121/117).
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- HF Nurse Up-titration: Intervention: The cardiologist prescribes drugs and, driven by protocol, the HF nurse implements the up-titration.
  HF nurse up-titration: Up-titration of Beta-Blocker (BB) in Heart Failure " De Novo" EF≤ 40% Patients. Protocol based on 2012 European Society of Cardiology (ESC) HF guidelines. Cardiologist prescription and support
  HF nurse up-titration: Up-titration of Angiotensin Converting Enzyme Inhibitor (ACEI) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 ESC HF guidelines. Cardiologist prescription and support
  HF nurse up-titration: Up-titration of Angiotensin II Receptor Blocker (ARB) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 ESC HF guidelines with cardiologist prescription and support
  HF nurse up-titration: Up-titration of Mineralocorticoid Receptor Antagonist (MRA) in Heart Failure " De Novo" EF≤ 40% patients. Protocol based on 2012 ESC HF guidelines. Cardiologist prescription and support
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 121 | 117
pg/ml | -1577 (3225) | -1593 (2733)
Statistical Analysis 1: Comparison: Heart Failure (HF) Cardiologist Up-titration vs HF Nurse Up-titration; Test type: Non-Inferiority — Equivalence margin of 5%; p = 0.97, t-test, 2 sided; Mean Difference (Final Values) = 16.47, 95% CI 2-sided [-781 to 748]

13. Secondary Outcome: 6 Minute Walking Test
Description: 6 minute walking test improvement ( change) meters.Improvement (difference of change from baseline to 6 months between groups Six minute walking test. Measurement of exercise capacity is an integral element in assessment of patients with cardiopulmonary disease. It provides information regarding functional capacity, response to therapy and prognosis across a range of chronic cardiopulmonary conditions. The six-minute walk test (6MWT) measures the distance (meters) an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 138 | 136
meters | 50.49 (74.20) | 57.76 (79.97)
Statistical Analysis 1: Comparison: Heart Failure (HF) Cardiologist Up-titration vs HF Nurse Up-titration; Test type: Non-Inferiority — Equivalence margin of 5%; p = 0.44, t-test, 2 sided; Mean Difference (Final Values) = 7.28, 95% CI 2-sided [-11.27 to 25.83]

14. Secondary Outcome: Number of Participants n(%) in New York Heart Association Functional Classification I,II,III,IV
Description: Number of participants class I-IV New York Heart Association (NYHA) functional classification, based on severity of symptoms and physical activity:
  NYHA I (better): No limitation of physical activity; NYHA II: Slight limitation of ordinary physical activity, breathlessness; NYHA III: marked limitation of physical activity. Comfortable at rest, but less than ordinary activity results in undue breathlessness, fatigue or palpitations; NYHA IV ( worse): unable to carry on any physical activity without discomfort.Symptoms at rest can be present. If any physical activity is undertaken discomfort is increased.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 137 | 135
Participants
  NYHA I | 47 | 59
  NYHA II | 86 | 72
  NYHA III | 4 | 4
  NYHA IV | 0 | 0

15. Secondary Outcome: Quality of Life: MLWHFQ
Description: Quality of Life, measured by Minnesota Living with Heart Failure Questionnaire. Improvement (change) from baseline to 6 months.
  Minnesota Living With Heart Failure Questionnaire (MLWHFQ). The content of this questionnaire was selected to be representative of the ways heart failure and treatments can affect the key physical, emotional, social and mental dimensions of quality of life of patients with heart failure. It consist of 21-items with score 0-5. Final evaluation moves from 0 (none) to 105 (very much); a lower score means better quality of life.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 138 | 136
score on a scale | -25.01 (23.22) | -26.37 (24.53)
Statistical Analysis 1: Comparison: Heart Failure (HF) Cardiologist Up-titration vs HF Nurse Up-titration; Test type: Non-Inferiority — Equivalence margin of 5%; p = 0.75, t-test, 2 sided; Mean Difference (Final Values) = -0.91, 95% CI 2-sided [-6.63 to 4.81]

16. Secondary Outcome: European Quality of Life Scale: EuroQol- 5 Dimension Index
Description: European Quality of Life Scale: EuroQol- 5 Dimension index (Range: 1 full health-0 death). It measures health status self-reported by the patient. It has 5 domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is divided into three levels: 1 no problem; 2 some or moderate problems; 3 extreme problems. The EuroQol Research Foundation converts this information into a single summary index, by applying a formula that attaches specific country values (called weights) to each of the levels in each dimension. The index is calculated by subtracting the mentioned weights from 1, the value for full health.
  We measured the EuroQol-5D index improvement (change) from baseline to 6 months.
  More information in: EQ-5D-3L-User-Guide_version-6.0 (1).pdf
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 138 | 136
score on a scale | 0.04 (0.28) | 0.08 (0.23)
Statistical Analysis 1: Comparison: Heart Failure (HF) Cardiologist Up-titration vs HF Nurse Up-titration; Test type: Non-Inferiority — Equivalence margin of 5%; p = 0.20, t-test, 2 sided; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.2 to 0.28]

17. Secondary Outcome: Number of Patients With Admissions Due to Heart Failure (HF)
Description: Number of patients with hospital admissions due to Heart Failure. From Baseline to 6 months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 145 | 144
Participants | 9 | 1
Statistical Analysis 1: Comparison: Heart Failure (HF) Cardiologist Up-titration vs HF Nurse Up-titration; Test type: Equivalence — equivalence margin of 5%; p = 0.01, Chi-squared; Difference in percentages = -5.5, 95% CI 2-sided [-9.7 to -1.4]

18. Secondary Outcome: Number of Patients With Deaths
Description: Number of Patients with deaths due to Cardiovascular and non cardiovascular causes
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 4 | 3
Participants
  mortality due to cardiovascular causes | 2 | 2
  mortality due to non cardiovascular causes | 2 | 1
Statistical Analysis 1: Comparison: Heart Failure (HF) Cardiologist Up-titration vs HF Nurse Up-titration; Test type: Non-Inferiority — Equivalence margin of 5%; p = 0.71, Chi-squared; Equivalence margin of 7%; Difference in percentages = -0.68, 95% CI 2-sided [-4.2 to 2.87]

19. Secondary Outcome: ACEI % Relative Dose (Mean) With Regard to Target Dose
Description: ACEI mean Relative dose is the mean dose of ACEI achieved 4 months after starting titration, relative to target dose (%) described in European guidelines
Time Frame: 4 Months
Measure: Mean (Standard Deviation); unit: percentage of target dose
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 115 | 115
percentage of target dose | 56.13 (30.4) | 72.61 (29.8)
Statistical Analysis 1: Comparison: Heart Failure (HF) Cardiologist Up-titration vs HF Nurse Up-titration; Test type: Non-Inferiority — Equivalence margin of 7%; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 16.5, 95% CI 2-sided [8.7 to 24.3]

20. Secondary Outcome: ARB % Relative Dose (Mean) With Regard to Target Dose
Description: ARB, angiotensin II receptor blockers, mean relative dose ( % to target dose). Target dose is described in European guidelines.
  Measured at 4 months after starting titration.
Time Frame: 4 months
Population: During the titration process several patients that at baseline did not have ARB prescription were prescribed this drug.
Measure: Mean (Standard Deviation); unit: percentage of target dose
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 20 | 18
percentage of target dose | 43.51 (33.7) | 44.48 (33.5)
Statistical Analysis 1: Comparison: Heart Failure (HF) Cardiologist Up-titration vs HF Nurse Up-titration; Test type: Non-Inferiority — Equivalence margin of 7%; p = 0.93, t-test, 2 sided; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-15.1 to 17.1]

21. Secondary Outcome: MRA % Relative Dose (Mean) With Regard to Target Dose
Description: MRA % relative dose (mean) is the mean dose achieved 4 months after starting titration with regard to target dose (%) described in european guidelines
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: percentage of target dose
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
Number analyzed (Participants) | 127 | 125
percentage of target dose | 70.47 (29.8) | 71.00 (32.1)
Statistical Analysis 1: Comparison: Heart Failure (HF) Cardiologist Up-titration vs HF Nurse Up-titration; Test type: Non-Inferiority — Equivalence margin of 7%; p = 0.86, t-test, 2 sided; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-7.1 to 8.2]

ADVERSE EVENTS:
Time Frame: From Baseline to 6 months
Arm/Group | Heart Failure (HF) Cardiologist Up-titration | HF Nurse Up-titration
All-Cause Mortality (participants affected / at risk) | 4/145 | 3/144
Serious Adverse Events (participants affected / at risk) | 11/145 | 2/144
Other Adverse Events (participants affected / at risk) | 20/145 | 22/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heart Failure (HF) Cardiologist Up-titration (N=145) | HF Nurse Up-titration (N=144)
hospitalizations due to cardiovascular cause (Cardiac disorders) | 11 (11) | 2 (2) — unplanned hospitalizations due to cardiovascular cause (not due to non cardiovascular cause)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Heart Failure (HF) Cardiologist Up-titration (N=145) | HF Nurse Up-titration (N=144)
heart rate <50 bpm (Cardiac disorders) | 7 (7) | 10 (10) — heart rate < 50 bpm, bradycardia possibly due to the titration process
symptomatic hypotension (Cardiac disorders) | 13 (13) | 12 (12) — symptomatic hypotension possibly due to the titration process

LIMITATIONS AND CAVEATS:
the implementation of ETIFIC in a single country; its recruitment characteristics, inclusion of de novo HF patients exclusively, relatively young patients and the low percentage of women and patients with ischemic heart disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-03-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT02546856/Prot_000.pdf
  • Statistical Analysis Plan (2015-03-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT02546856/SAP_001.pdf